CLINICAL TRIAL: NCT07299227
Title: Impact of Balloon Pulmonary Angioplasty in CTEPH on Cardiac and Pulmonary Physiology as Assessed by State-of-the-art Cardiovascular Magnetic Resonance 4D Flow Haemodynamics
Brief Title: Impact of BPA in CTEPH on Cardiac and Pulmonary Physiology Assessed by CMR-derived 4D Flow Haemodynamics
Status: Recruiting | Type: Observational
Sponsor: Kerckhoff Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: AZ 158/24
Record Dates: First submitted 2025-08-27; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: CTEPH
Keywords: CTEPH; CMR; 4D flow

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CTEPH patient

SUMMARY:
Patients with CTEPH referred for evaluation and conduction of BPA undergo standard of care diagnostic tests and treatment. This includes conventional echocardiographic, RHC and non-invasive (CT/CMR) or invasive (coronary angiography) coronary artery disease work-up. BPA will be conducted in generally 5 to 6 consecutive sessions. CMR will be performed prior to first and following the last intervention. Patient recruitment will be performed within 3 years, that is the last BPA session of the last patient in will have been performed at 3 years time.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to BPA
* clinical indication for CMR
* capability to give informed consent

Exclusion Criteria:

* general: non-compliance, <18 years of age, pregnancy
* contraindications for CMR (non-CMR compatible device, chronic kidney disease (eGFR <30ml/min), allergies (medications)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All CTEPH patients to undergo BPA
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  1a) Changes in right cardiac function (RV EF %)
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  1b) Changes in cardiac function (RV GLS%)
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  2a) Changes in pulmonary artery flow (peak flow m/s)
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  2b) Changes in pulmonary artery flow (mean flow m/s)
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  2c) Changes in pulmonary artery flow (pulse wave velocity m/s)

SECONDARY OUTCOMES:
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  1a) Change in LV tissue composition - T1 (ms)
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  1b) Change in LV tissue composition - ECV (%)
Impact of BPA on cardio-pulmonary vascular physiology | 1 year
  2) Change in RA phasic function (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Kerckhoff-Klinik, Bad Nauheim, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Undecided